CLINICAL TRIAL: NCT06989723
Title: Evaluation of Pioglitazone and Empagliflozin Combination Therapy in Type 2 Diabetes Patients With Metabolic Dysfunction-Associated Fatty Liver Disease
Brief Title: Pioglitazone and Empagliflozin for Fatty Liver Disease in Type 2 Diabetes
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: Celltrion (Industry)
Responsible Party: Principal Investigator, Soo Lim, Clinical Professor and Principal Investigator, Division of Endocrinology, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B-2407-911-001
Record Dates: First submitted 2025-04-29; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Type 2 Diabetes; Fatty Liver
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Fatty Liver | interventions — Pioglitazone; empagliflozin

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: A randomization sequence will be generated prior to patient enrollment. Patients will be enrolled before the treatment allocation is disclosed. The allocation sequence will be revealed at the time of group assignment, after which the prescribed intervention will be administered. Until group assignment, both the enrolling investigators and the patients who have provided informed consent will remain unaware of the assigned treatment group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pioglitazone (Experimental): Pioglitazone 15mg
  Interventions: Drug: Empagliflozin 10 MG [Jardiance]
- Empagliflozin (Experimental): Empagliflozin 10mg
  Interventions: Drug: Pioglitazone 15 MG [Actos]
- Pioglitazone & Empagliflozin (Experimental): Pioglitazone 15mg + Empagliflozin 10mg
  Interventions: Drug: Empagliflozin 10 MG [Jardiance] + Pioglitazone 15 MG [Actos]

INTERVENTIONS:
Drug: Pioglitazone 15 MG [Actos] — Participants will receive pioglitazone 15 mg, administered orally once daily. The tablet may be taken with or without food.
  Arms: Empagliflozin
Drug: Empagliflozin 10 MG [Jardiance] — Participants will receive empagliflozin 10 mg, administered orally once daily. The tablet may be taken with or without food.
  Arms: Pioglitazone
Drug: Empagliflozin 10 MG [Jardiance] + Pioglitazone 15 MG [Actos] — Participants will receive one tablet of pioglitazone 15 mg and one tablet of empagliflozin 10 mg, administered orally once daily. Both tablets may be taken with or without food.
  Arms: Pioglitazone & Empagliflozin

SUMMARY:
This exploratory study will assess the efficacy of combined pioglitazone and empagliflozin therapy in improving hepatic and metabolic outcomes in patients with type 2 diabetes mellitus and metabolic dysfunction-associated fatty liver disease (MAFLD). Although each agent has shown beneficial effects individually, evidence on their combined impact on liver health is scarce. This study seeks to determine whether the combination therapy yields additive improvements in hepatic steatosis, inflammation, and fibrosis, potentially offering a new therapeutic strategy for diabetic patients with fatty liver disease.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 20 years or older.
2. Patients with inadequately controlled type 2 diabetes mellitus, defined as HbA1c between 7% and 10%, who are currently treated with either:

   * Combination therapy of metformin and a sulfonylurea, or
   * Combination therapy of metformin and a DPP-4 inhibitor, or
   * Metformin monotherapy, or
   * Triple therapy (including metformin) provided that sulfonylurea will be discontinued upon study enrollment.
3. Evidence of hepatic steatosis within the past 3 months, confirmed by Fibroscan with a controlled attenuation parameter (CAP) ≥ 268 dB/m (consistent with S2 or greater [≥10% hepatocyte steatosis] according to the 2024 EASL-EASD-EASO guidelines).
4. Presence of at least one of the following metabolic abnormalities:

   * Waist circumference ≥90 cm for men or ≥85 cm for women.
   * Blood pressure ≥130 mmHg systolic or ≥85 mmHg diastolic, or use of antihypertensive medication.
   * Serum triglycerides ≥150 mg/dL or current use of lipid-lowering agents.
   * HDL-cholesterol ≤45 mg/dL for men or ≤50 mg/dL for women.
   * HOMA-IR (Homeostatic Model Assessment of Insulin Resistance) ≥2.5.
   * Serum C-reactive protein (CRP) ≥2 mg/L.
5. No changes in anti-diabetic or metabolic medications within the past 3 months, unless the changes are deemed by the investigator not to affect study outcomes.

Exclusion Criteria:

1. Patients receiving insulin therapy or diagnosed with type 1 diabetes mellitus.
2. Use of the following medications within the past 3 months: GLP-1 receptor agonists, SGLT2 inhibitors, rosiglitazone (TZD), vitamin E, or ursodeoxycholic acid (UDCA).
3. Presence of secondary causes of hepatic steatosis unrelated to metabolic dysfunction, such as hepatitis B, hepatitis C, or alcoholic fatty liver disease.
4. Use of medications known to induce hepatic steatosis, including valproic acid, estrogen, tamoxifen, amiodarone, or chloroquine.
5. Severe organ failure, defined as:

   * Liver failure: AST or ALT > 5 times the upper normal limit (UNL), serum albumin < 3.2 g/dL, platelet count < 60,000/µL, or Child-Pugh-Turcotte stage B or C.
   * Renal failure: Serum creatinine ≥ 2.0 mg/dL, estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73 m² (CKD-EPI formula), or patients with end-stage renal disease or on dialysis.
6. Presence of hepatocellular carcinoma, active malignancy, or metastatic cancer.
7. History of or active bladder cancer.
8. History of heart failure or current diagnosis of heart failure.
9. Presence of terminal illnesses.
10. History of gallstone disease, chronic pancreatitis, or acute pancreatitis.
11. Underweight patients (body mass index [BMI] < 18.5 kg/m²).
12. Pregnant women or women planning to become pregnant.
13. Known hypersensitivity to the active ingredients or excipients of the study medications.
14. History of diabetic ketoacidosis.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants Achieving HbA1c Treatment Targets | 24 weeks
  Percentage of participants who achieve the predefined HbA1c treatment goal at 24 weeks.
Change in Fibroscan Controlled Attenuation Parameter (CAP) Score | 24 weeks
  Assessment of changes in hepatic steatosis as measured by the controlled attenuation parameter (CAP) score using Fibroscan technology over a 24-week period.

SECONDARY OUTCOMES:
Change in HbA1c Levels | 24 weeks
  Change in glycated hemoglobin (HbA1c) from baseline after 24 weeks of treatment.
Change in Liver Stiffness Measurement | 24 weeks
  Change in liver stiffness measurement (LSM) assessed using Fibroscan
Change in Non-Invasive Blood-Based Fibrosis Markers | 12 weeks, 24 weeks
  Change in NAFLD score, Fibrosis-4 (FIB-4) index, and AST to Platelet Ratio Index (APRI) over 12 and 24 weeks.
Change in Anthropometric Measures | 12 weeks, 24 weeks
  Changes in metabolic parameters including body weight, body mass index (BMI), waist circumference
Change in Lipid Parameters | 12 weeks, 24 weeks
  Changes in blood lipid profile (total cholesterol, LDL-c, HDL-c, triglycerides)
Change in Liver Function Tests | 12 weeks, 24 weeks
  Change in liver function markers including AST, ALT, gamma-glutamyl transferase (gamma-GT), albumin, bilirubin, and prothrombin time
Change in Fibrosis Biomarker | 12 weeks, 24 weeks
  Change in serum type IV collagen levels
Change in Inflammatory Biomarker | 12 weeks, 24 weeks
  Change in high-sensitivity C-reactive protein (hs-CRP) levels

OTHER OUTCOMES:
Change in Other Blood Biomarkers | 24 weeks
  Change in ketone body levels
Change in Proteinuria | 24 weeks
  Change in urinary albumin-to-creatinine ratio, protein-to-creatinine ratio

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, South Korea

IPD SHARING:
Plan to Share IPD: Undecided